CLINICAL TRIAL: NCT04206904
Title: Prevalence of Frailty in Patients With a Cardiovascular Disease and Correlations With Markers of Exercise
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Invesigator, Hasselt University
Other Study IDs: FrCR
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Frailty
Keywords: older adults; cardiovascular diseases; maximal exercise test
MeSH Terms: conditions — Frailty; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the first part of this study the prevalence of frailty in patients with cardiovascular disease will be examined. Frailty is defined as a progressive age-related decline in physiological systems that results in decreased reserves of intrinsic capacity, which confers extreme vulnerability to stressors. Patients (≥65 years, men and women) suffering from heart failure or undergoing a coronary artery bypass grafing (CABG) or percutaneous coronary intervention (PCI) will be included. Based on the phenotype of Fried, frailty will be examined in the physical domain. Moreover, the nutritional, social, psychological and cognitive domain of frailty will be examined. This will result in a total score of 0 (no frailty) to 24 (severe frailty), divided into four categories: no frailty (score 0-6), minor frailty (score 7-12), moderate frailty (score 13-18) or severe frailty (score 18-24).

Besides this frailty protocol, a few other measurements will be completed to collect additional information about the functioning of the patient.

At discharge from the hospital, some of these patients will start with a cardiac rehabilitation program. To define the exercise intensity of this program, patients will perform a maximal exercise test (CPET). In the second part of this study, correlations will be examined between markers of frailty and markers of exercise from the CPET (e.g. maximal heart rate, maximal oxygen uptake).

ELIGIBILITY:
Inclusion Criteria:

Men and women with an age of at least 65 years at the start of the study; Staying in Jessa Hospital for PCI, CABG or heart failure

Exclusion Criteria:

A persistently unstable clinical condition at baseline visit (angina, advanced conduction disturbances, threatening ventricular arrhythmias, acute heart failure, clinical condition requiring interventions such as acute renal failure, Hb <9,0 mg/dl, presence of end-stage disease or the lack of informed consent to study participation)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women with an age of at least 65 years at the start of the study who are admitted to Jessa Hospital Hasselt because of suffering from coronary artery diseases (with planned PCI or CABG surgery) or heart failure
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Level of (in)dependence via the Katz scale | At baseline
  Evaluation of the level of (in)dependence in activities of daily life via a 4-point scale (1-4)
Nutritional status via the Mini Nutritional Assessment (MNA) | At baseline
  Examination of the nutritional status of the patient via a questionnaire (30 points)
Level of physical activity via the International Physical Activity Questionnaire (IPAQ) | At baseline
  Examination of the level of physical activity of the patient via a questionnaire
Cognitive status via the Mini Mental State Examination (MMSE) | At baseline
  Examination of the cognitive status of the patient via a short screening (30 points)
Psychological status via the Geriatric Depression Scale (GDS-15) | At baseline
  Examination of the presence/absence of a depressive mood via a questionnaire (15 questions/15 points)
Concern about falling via the Falls Efficacy Scale (FES-I) | At baseline
  Examination of the level of concern about falling during social and physical activities via a questionnaire (16 questions/ 64 points)
Weight loss via the evaluation of body weight | At baseline
  Evaluation of involuntary loss of body weight in the previous months
Gait speed via the 4.6 meter walking test | At baseline
  Examination of the walking speed of the patient
Evaluation of handgrip strength | At baseline
  Evaluation of the handgrip strength of the patient via handheld dynamometry
Examination of mobility/balance/muscle strength/risk of falling via the Timed Up and Go Test (TUG) | At baseline
  The Timed Up and Go Test measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. By combining this test with a motor or cognitive dual task, the risk of falling of the patient will be examined.
Comorbidities via the record of medication use | At baseline
  Record of cardiac and other medications
Evaluation of lower limb strength | At baseline
  Evaluation of lower limb strength of the patient via Microfet measurements
Evaluation of functional lower limb strength | At baseline
  Evaluation of functional lower limb strength of the patient via the Timed Chair Stand Test

SECONDARY OUTCOMES:
Correlations between frailty (via the primary frailty outcome measures) and exercise parameters (via the maximal exercise test (CPET) | At the start of the cardiac rehabilitation program
  Evaluation of correlations between frailty characteristics (from the primary outcome measures) and exercise parameters from a maximal exercise test (CPET) (performed at the start of a cardiac rehabilitation program).

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital Campus Virga Jesse, Hasselt, Limburg, Belgium